CLINICAL TRIAL: NCT00451568
Title: Metformin and Oral Contraceptives in PCOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Marianne Andersen, Professor, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 027
Record Dates: First submitted 2007-03-22; First posted 2007-03-23 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic ovary syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): metformin
  Interventions: Drug: Metformin
- 2 (Active Comparator): desorelle
  Interventions: Drug: Desorelle
- 3 (Active Comparator): desorelle + metformin
  Interventions: Drug: Metformin; Drug: Desorelle

INTERVENTIONS:
Drug: Metformin — 500 mg 2 tablets 2 times a day
  Arms: 1; 3
Drug: Desorelle — 1 tablet/day in 21 days
  Arms: 2; 3

SUMMARY:
Background: PCOS is a common condition with a prevalence of 5-8 % in premenopausal women. More than 50% of PCOS patients are insulin resistant and have a diabetes risk 5-8 times higher than age- and weight-matched controls. Studies using insulin sensitizers in PCOS found increased insulin sensitivity and decreased insulin levels to be followed by decreased androgen levels and improved ovulatory function. No studies however, evaluated the long term effects of insulin sensitizing treatment.

Oral contraceptives normalize menstrual cycles and suppress androgen levels in PCOS, however no long-term studies evaluated the effects of combined treatment with metformin and oral contraceptives in PCOS.

Design: Randomized open study in 3*30 PCOS patients. Patients are randomised to 24 months of treatment with 1: metformin, 2: metformin and oral contraceptives or 3: oral contraceptives.

Primary outcome measures: fasting insulin, AUC insulin. Secundary endpoints: BMI, WHR, LH, FSH, total and free-testosterone, c-peptid, urinary cortisol, AUC for insulin, glucose and c-peptid during OGTT.

Inclusioncriteria:

1. Irregular menses or anovulaty cycles
2. High free testosterone > 0,035 nmol/l or hirsutism
3. PCO in vaginal US Criteria 1 and 2 OR 2 and 3.

Design:

DETAILED DESCRIPTION:
90 patients are included and randomized to 12 months of treatment with metformin (1000+1000 mg/d) or OCP (150 mg desogestrel 30 microgram ethinylestradiol) or combined treatment (metformin+OCP).

Patients attend a biochemical and physical examination at study inclusion and at 12 months. Patients attend for registration of side effects and compliance after 6 months of study duration. Safety tests are performed at all three visits and include weight, blood pressure, HbA1c, liver enzymes, electrolytes, and white blood cell count. Pregnancy tests are performed by the participants each month. Patients are given general advice on lifestyle intervention. Patients are excluded if they initiated medical treatment with possible hormonal and metabolic effects during the intervention period. Lifestyle intervention is allowed. Laser treatment is offered to patients with moderate or severe facial hirsutism and patients are allowed to shave/wax. The patients accept not applying cosmetic treatment 3-4 days before attending for evaluation at the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Irregular menses or anovulaty cycles
* High free testosterone > 0.035 nmol/l or hirsutism
* PCO in vaginal US Criteria 1 and 2 OR 2 and 3

Exclusion Criteria:

* Age > 18 years
* Postmenopausal
* Diagnosis diabetes mellitus
* Use of medicine known to affect hormones measured in the project
* Pregnancy or planned pregnancy during study period
* Non-Caucasian
* Previous tromboembolic disease
* Heavy smoker > 35 years and BMI > 35 kg/m2

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2007-03; Primary Completion 2012-01 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Changes in fasting insulin and area under the curve for insulin (2 hours) | 12 months

SECONDARY OUTCOMES:
Changes in BMD, BMI, WHR, LH, FSH, total and free testosterone, fasting blood glucose, fasting C-peptide, urine-cortisol secretion, body composition, number of hypoglycaemic cases, AUC for insulin, glucose and C-peptide during OGTT (2 and 5 ho | 12 months
Changes in cortisol metabolism | 12 months
Changes in the prevalence of reactive hypoglycemia and areal under the curve for glucose (5 hours) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Andersen, MD, PhD, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

REFERENCES:
- [Derived] Glintborg D, Petersen MH, Ravn P, Hermann AP, Andersen M. Comparison of regional fat mass measurement by whole body DXA scans and anthropometric measures to predict insulin resistance in women with polycystic ovary syndrome and controls. Acta Obstet Gynecol Scand. 2016 Nov;95(11):1235-1243. doi: 10.1111/aogs.12964. PMID 27529295
- [Derived] Mumm H, Altinok ML, Henriksen JE, Ravn P, Glintborg D, Andersen M. Prevalence and possible mechanisms of reactive hypoglycemia in polycystic ovary syndrome. Hum Reprod. 2016 May;31(5):1105-12. doi: 10.1093/humrep/dew046. Epub 2016 Mar 23. PMID 27008892
- [Derived] Glintborg D, Mumm H, Altinok ML, Richelsen B, Bruun JM, Andersen M. Adiponectin, interleukin-6, monocyte chemoattractant protein-1, and regional fat mass during 12-month randomized treatment with metformin and/or oral contraceptives in polycystic ovary syndrome. J Endocrinol Invest. 2014 Aug;37(8):757-764. doi: 10.1007/s40618-014-0103-8. Epub 2014 Jun 7. PMID 24906976
- [Derived] Glintborg D, Altinok ML, Mumm H, Hermann AP, Ravn P, Andersen M. Body composition is improved during 12 months' treatment with metformin alone or combined with oral contraceptives compared with treatment with oral contraceptives in polycystic ovary syndrome. J Clin Endocrinol Metab. 2014 Jul;99(7):2584-91. doi: 10.1210/jc.2014-1135. Epub 2014 Apr 17. PMID 24742124